CLINICAL TRIAL: NCT03571308
Title: A Phase Ib/II Combination of Acalabrutinib With R-CHOP for Patient Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Combination of Acalabrutinib With R-CHOP for Patient Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: ACCEPT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RHM CAN 1129
Record Dates: First submitted 2017-10-06; First posted 2018-06-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Diffused Large B-Cell Lymphoma; Acalabrunitib; Bruton Tyrosine Kinase; R-CHOP; Molecular Profiling; Chemoimmunotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — acalabrutinib; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisolone

STUDY DESIGN:
Masking Description: A multicentre open-label non-randomised phase Ib/II two stage trial. Stage 1 - dose escalation will proceed until a maximum tolerated dose (MTD) is defined or the maximal administered dose (MAD) is determined in order to define the recommended Phase II dose (RP2D). 6 - 24 patients. Stage 2 - expansion to gain additional information on safety and efficacy at the RP2D from a total of 15 patients recruited.
  Patients will receive conventionally dosed R-CHOP chemotherapy for 6 cycles with acalabrutinib introduced on cycle 2 onwards, at a dosage according to cohort number. This will allow for both clarity in the toxicity profile of the combination and also assess the impact of acalabrutinib on ADCC.
  patients who do not complete six cycles of treatment for reasons other than toxicity will be replaced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CHOP + Acalabrutinib (Experimental): Open-label non-randomised phase Ib/II study conducted in two stages. Phase I will see two doses of acalabrutinib tested. R-CHOP + acalabrutinib will be given for 6 cycles on a 21 day cycle and then two cycles of acalabrutinib only for a total of 56 days. Acalabrutinib will be introduced at Cycle 2.
  Phase II will see the recommended phase 2 dose used on the same treatment regimen.
  Interventions: Drug: R-CHOP + acalabrutinib

INTERVENTIONS:
Drug: R-CHOP + acalabrutinib — Patient will be given R-CHOP and acalabrutinib
  Other Names: Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisolone; Acalabrutinib

SUMMARY:
Previously untreated CD20 positive diffuse large B-cell lymphoma (DLBCL) requiring full course chemoimmunotherapy.

DETAILED DESCRIPTION:
Open-label non-randomised phase Ib/II study conducted in two stages. Stage 1 will be dose escalation in a modified classical 6+6 design. Stage 2 will be an expansion cohort to gain additional information on safety and efficacy at the recommended phase II dose of acalabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL, expressing CD20. Sufficient diagnostic material should be available to forward to a central laboratory for gene expression profiling and pathology review.
* Measurable disease of at least 15mm.
* Not previously treated for lymphoma and fit enough to receive combination chemoimmunotherapy with curative intent.
* Stage IAX (bulk defined as lymph node diameter >10cm) to stage IV disease and deemed to require a full course of chemotherapy. Patients with non-bulky IE disease will not be eligible.
* ECOG performance status 0-2 or 3 if this is directly attributable to lymphoma.
* Adequate bone marrow function with platelets > 100x109/L; neutrophils > 1.0x109/L at study entry, unless lower figures are attributable to lymphoma.
* Measured or calculated creatinine clearance > 30mls/min, (calculated using the formula of Cockcroft and Gault [(140-Age) x Mass (kg) x (1.04 (for women) or 1.23 (for men))/Serum Creatinine (µmolL)].
* Serum bilirubin < 35μmol/L and transaminases < 2.5x upper limit of normal at time of study entry
* Cardiac function sufficient to tolerate 300mg/m2 of doxorubicin. A pre-treatment echocardiogram or MUGA is required to establish baseline LVEF equal to or greater than 55%.
* No concurrent uncontrolled medical condition.
* Life expectancy > 3 months.
* Aged 16 years or above.
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent.

Exclusion Criteria:

Patients will be excluded from the study entry if any of the following criteria are met:

* Previous history of treated or untreated indolent lymphoma. However newly diagnosed patients with DLBCL who are found to also have small cell infiltration of the bone marrow or other diagnostic material (discordant lymphoma) will be eligible.
* Patients who have received immunisation with a live vaccine within four weeks prior to enrolment will be ineligible.
* Diagnosis of primary mediastinal lymphoma.
* Diagnosis of primary Central Nervous System lymphoma.
* History of stroke or intracranial haemorrhage in preceding 6 months.
* History of bleeding diathesis (eg, haemophilia, von Willebrand disease).
* Requires or receiving anticoagulation with warfarin or equivalent antagonists (eg, phenprocoumon) within 7 days of first dose of acalabrutinib. However patients using therapeutic low molecule weight heparin or low dose aspirin will be eligible.
* Prior exposure to a BCR inhibitor (eg, Btk inhibitors, phosphoinositide-3 kinase (PI3K), or Syk inhibitors) or BCL-2 inhibitor (eg, ABT-199)
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
* Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Patients receiving proton pump inhibitors who switch to short-acting H2-receptor antagonists or antacids are eligible for enrolment into this study.
* Uncontrolled systemic infection.
* Major surgery in the preceding 4 weeks of first dose of study drug. If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec at screening.
* Serological positivity for Hepatitis B, C, or known HIV infection. As per standard of care, prior to initiation of immunochemotherapy, the results of hepatitis serology should be known prior to commencement of therapy.

  * Positive test results for chronic HBV infection (defined as positive HBsAg serology) will not be eligible. Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) will not be eligible. Patients who have protective titres of hepatitis B surface antibody (HBsAb) after vaccination will be eligible.
  * Positive test results for hepatitis C (HCV antibody serology testing) will not be eligible.
* Women who are sexually active and can bear children must agree to use highly effective forms of contraception or abstinence during the study and for 12 months after the last treatment dose. Highly effective forms of contraception are defined in Section 4.7.
* Breastfeeding or pregnant women.
* Men who are sexually active and can father children must agree to use highly effective forms of contraception or abstinence during the study and for 12 months after the last treatment dose. Highly effective forms of contraception are defined in Section 4.7.
* Men must agree to refrain from sperm donation during the study and for 12 months after the last treatment dose.
* Serious medical or psychiatric illness likely to affect participation or that may compromise the ability to give informed consent.
* Prior malignancy (other than DLBCL), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years. Note: these cases must be discussed with SCTU.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, gastric bypass, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction or gastric restrictions and bariatric surgery, such as gastric bypass.
* Any immunotherapy within 4 weeks of 1st dose of the study.
* Concurrent participation in another therapeutic clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose limiting toxicity of acalabrutinib combined to R-CHOP | 18 months
  Define recommended dose for Phase II evaluation of acalabrutinib with R-CHOP examining safety and toxicity of combination
Phase II: Overall response rate of the combination acalabrutinib and R-CHOP | 36 months
  Document anti-tumour activity of acalabrutinb in combination wit R-CHOP in patients with previously untreated CD20 positive DLBCL
Safety of the combination acalabrutinib and R-CHOP as determined by treatment-related adverse events as assessed by CTCAE v4.03. | 12 months
  To determine additional safety information of acalabrutinib in combination with R-CHOP by treatment-related adverse events as assessed by CTCAE v4.03.

SECONDARY OUTCOMES:
Pharmacokinetics of acalabrutinib using area under the plasma concentration versus time curve (AUC) | 24 months
  To determine the pharmacokinetic (PK) profile of acalabrutinib when given in combination with R-CHOP in patients with DLBCL
Maximum Plasma Concentration (Cmax) of acalabrutinib | 24 months
  To determine the pharmacokinetic (PK) profile of acalabrutinib when given in combination with R-CHOP in patients with DLBCLPK parameter.
Time after administration when maximum concentration of acalabrutinib in the plasma is reached (Tmax) | 24 months
  To determine the pharmacokinetic (PK) profile of acalabrutinib when given in combination with R-CHOP in patients with DLBCL
Time required for concentration of acalabrutinib to reach half original value (T1/2) | 24 months
  To determine the pharmacokinetic (PK) profile of acalabrutinib when given in combination with R-CHOP in patients with DLBCL
Overall response rate of the combination acalabrutinib and R-CHOP according to cell of origin. | 24 months
  To evaluate the effect of acalabrutinib in combination with R-CHOP on outcomes according to cell of origin
Two years progression-free survival | 24 months
  To measure the duration of response to acalabrutinib in combination with R-CHOP over a follow-up period of 2 years
Two years overall survival | 24 months
  To measure the duration of response to acalabrutinib in combination with R-CHOP over a follow-up period of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andy Davies, Principal Investigator — Southampton University Hospital NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Southampton University Hospitals NHS Tust, Southampton, Hampshire
  - St James's University Hospital, Leeds
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital Campus, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ASH 62nd Annual Meeting 2020 abstract — https://ash.confex.com/ash/2020/webprogram/Paper134546.html